CLINICAL TRIAL: NCT04834193
Title: Wet-suction Versus Slow-pull Technique for Endoscopic Ultrasound-guided Fine-needle Biopsy of Solid Lesions: a Multicentric Randomized Controlled Trial
Brief Title: Wet-suction Versus Slow-pull for EUS-FNB of Solid Lesions
Acronym: WEST-FNB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Stefano Francesco Crinò, MD, Principal Investigator, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 18/22.09.2020
Record Dates: First submitted 2021-03-29; First posted 2021-04-08 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Endoscopic Ultrasound; Fine-needle Aspiration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WET-SUCTION (Experimental): The stylet will be removed and the needle will be pre-flushed with 1-2mL of saline. The lesion will then be punctured, and suction will be applied using a 10-mL pre-vacuum syringe. The sample collected will be pushed into a formalin vial with saline.
  Interventions: Procedure: Endoscopic ultrasound-guided fine-needle biopsy
- SLOW-PULL (Active Comparator): After puncturing the lesion, the stylet will be slowly and gradually withdrawn for at least 40cm. The sample will be pushed into formalin using the stylet.
  Interventions: Procedure: Endoscopic ultrasound-guided fine-needle biopsy

INTERVENTIONS:
Procedure: Endoscopic ultrasound-guided fine-needle biopsy — Solid lesions will be sampled under endoscopic ultrasound guidance using the two techniques (wet-suction and slow-pull)

SUMMARY:
A randomized cross-over study investigating the impact of two different suction techniques on histological yield and sample quality of specimens collected by endoscopic ultrasound biopsy from solid lesions using histology needles.

ELIGIBILITY:
Inclusion Criteria:

* Solid pancreatic lesions 3 1cm
* Peri-GI tract lymph nodes 3 1cm
* Peri-GI tract masses
* Lesions of the GI wall
* Signed informed consent

Exclusion Criteria:

* Pancreatic cystic lesions (more than 50% of the volume)
* Diameter of lesion ≤ 1 cm
* Lesion not seen at EUS
* Pregnancy
* Coagulopathy (platelet count <50.000/mm3 and/or international normalized ratio >1.5);
* Severe cardiorespiratory dysfunction precluding endoscopy;
* Failure to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Histologic yield | 6 months
  The rate of samples containing a tissue "core" (yes/no) for histological evaluation, defined as an intact piece of tissue of at least 550 μ

SECONDARY OUTCOMES:
Tissue integrity | 6 months
  Tissue integrity will be evaluated by attributing a score from zero to 3 (3 represents the better outcome), according to the following score system:
  0: No cells/tissue
  1. Cytological specimen (disaggregated cells representative of the target lesion not allowing for tissue architectural assessment)
  2. Histologic microfragments (sample adequate for histological evaluation, namely an architecturally intact piece of tissue but without a "core")
  3. Histologic "core" (defined as an architecturally intact piece of tissue measuring at least 550 μ)
Blood contamination | 6 months
  Blood contamination will be evaluated by attributing a score from zero to 3 (3 represents the better outcome), according to the following score system:
  0: Only blood
  1. High blood contamination (>50% of the surface)
  2. Moderate blood contamination (25-50% of the surface)
  3. Low blood contamination (<25% of the surface)
Tumor fraction | 6 months
  The rate of samples containing an adequate tumor fraction ≥20 percent (i.e., ≥ 20 percent tumor cells in a background of benign nucleated cells).
Diagnostic accuracy | 6 months
  Diagnostic accuracy (defined as the ratio between the sum of true positive and true negative values divided by the number of lesions) will be calculated for each study arm

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Integrata Verona, Verona, Italy

REFERENCES:
- [Derived] Crino SF, Conti Bellocchi MC, Di Mitri R, Inzani F, Rimbas M, Lisotti A, Manfredi G, Teoh AYB, Mangiavillano B, Sendino O, Bernardoni L, Manfrin E, Scimeca D, Unti E, Carlino A, Voiosu T, Mateescu RB, Fusaroli P, Lega S, Buscarini E, Pergola L, Chan SM, Lamonaca L, Gines A, Fernandez-Esparrach G, Facciorusso A, Larghi A. Wet-suction versus slow-pull technique for endoscopic ultrasound-guided fine-needle biopsy: a multicenter, randomized, crossover trial. Endoscopy. 2023 Mar;55(3):225-234. doi: 10.1055/a-1915-1812. Epub 2022 Aug 1. PMID 35915956

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT04834193/Prot_SAP_000.pdf